CLINICAL TRIAL: NCT06126484
Title: Outcomes of Transcatheter Cardiac Interventions in Neonates With Congenital Heart Disease at Sohag University Hospital
Brief Title: Neonatal Transcatheter Cardiac Interventions at Sohag University Hospital
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Somia Sabry Mahmoud, Assistant lecturer of Pediatrics, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-10-04MD
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Transcatheter Neonatal Cardiac Interventions
Keywords: Catheter, neonates, congenital heart disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neonates with congenital heart disease (Other): Neonates with critical congenital heart diseases that require early catheter intervention
  Interventions: Procedure: transcatheter cardiac intervention

INTERVENTIONS:
Procedure: transcatheter cardiac intervention — Balloon atrial septostomy, PDA stent implantation, Pulmonary valvuloplasty, Aortic valvuloplasty, Balloon angioplasty of coarctation, PDA closure in preterm neonates

SUMMARY:
This study is performed to assess the safety, efficacy and outcome of transcatheter cardiac interventions in neonates with critical congenital heart disease at Sohag University Hospital

DETAILED DESCRIPTION:
This study includes neonates with critical congenital heart diseases that require early interventions Patients with untreated sepsis and coagulopathy are excluded.

Methods:

A) Clinical data: age, body weight and oxygen saturation B) Echocardiographic data: cardiac anatomical diagnosis. C) Catheterization data: vascular access, description of the defects, type of the device used, fluoroscopy time, radiation time, related complications and added interventions in the same setting.

D) Procedural details:

* All procedures will be performed under general anesthesia. procedures will be performed are;

  1. Balloon atrial septostomy.
  2. PDA stent implantation.
  3. Pulmonary valvuloplasty.
  4. Aortic valvuloplasty.
  5. Balloon angioplasty of coarctation.
  6. PDA device closure for preterm neonates.

     E) Post-procedure details:
* All the patients will be transferred to NICU.
* Prophylactic antibiotic therapy will be given to all patients.
* In patients with PDA stent; heparin infusion will be maintained for at least for 24-48 hours then acetylsalicylic acid: Dose; 5mg/kg/day will be added when oral feeding could be established until undergoing second-stage palliation or repair.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with critical congenital heart diseases that require early intervention

Exclusion Criteria:

* Untreated sepsis and coagulopathy.

Ages: 1 Hour to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
procedure related complications | 1 day
  complications that may occur during or after procedure

SECONDARY OUTCOMES:
Postprocedure NICU admission | 2 weeks
  complications after procedure in NICU

CONTACTS AND LOCATIONS:
Overall Officials: Somaia S Mahmoud, Master, Principal Investigator — Faculty of Medicine, Sohag University
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No